CLINICAL TRIAL: NCT05078372
Title: Comparison of the Effectiveness of the Use of Ropivacaine and Midazolam by Intraarticular vs Epidural Administration on Post-operative Analgesia After Isolated Arthroscopic ACL Reconstruction With Hamstring Autograft.
Brief Title: Ropivacaine and Midazolam by Intraarticular vs Epidural Administration in Arthroscopic ACL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Rodolfo Morales Avalos, MD, MSc, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN19-00003
Record Dates: First submitted 2021-09-19; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Anesthesia Injection Site; Knee Injuries
Keywords: Knee infiltration; Anterior Cruciate Ligament; Hamstring; Ropivacaine; Midazolam
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Two study groups will be generated, each consisting of 54 research subjects, randomly each recipient will receive epidural anesthesia with or without intraarticular ropivacaine. The group to which the patient belongs will be assigned through a computer program, the patient will not know to which group he belongs or what medication he will receive. The patients will be extracted from the external traumatology clinic
Who Masked: Participant, Investigator
Masking Description: Prior to being included in the study, the patient will be mentioned the times when he will receive the medication as well as the dosage of administration. The patient will not know what medication is being administered to him / her. The drug will be given to the anesthesist in unlabeled syringes without access to any information legend. In the same way, the study group only will be know by a doctor outside the research protocol and will not participate in any other phase of the study so that no member of the research team will know what medication was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine and midazolam epidural administration (Active Comparator): An elastomeric pump was prepared for epidural infusion. This was prepared with 150 mg (20 ml) of 0.75% ropivacaine plus midazolam at 50 mcg / kg / 12 hrs. The solution was made up to 125 ml with physiological solution.
  And 20 ml of physiological solution, was intraarticular administered as placebo.
  Interventions: Drug: ropivacaine and midazolam epidural administration
- Ropivacaine and midazolam intraarticular administration (Active Comparator): Ropivacaine 0.75% at 1.5 mg / kg was used with midazolam at 50 mcg / kg, to complete 20 ml of solution and was administrated on the knee articulation after tourniquet release.
  And an elastomeric pump was prepared for epidural infusion, with 150 ml of physiological solution as placebo.
  Interventions: Drug: ropivacaine and midazolam intraarticular administration

INTERVENTIONS:
Drug: ropivacaine and midazolam intraarticular administration — Patients undergoing ACL reconstruction with hamstring autograft who will receive ropivacaine and midazolam epidural administration for anesthesic technique for the procedure, and intraarticular administration of those drugs.
  Other Names: Ropiconest®; Ralecum®
  Arms: Ropivacaine and midazolam intraarticular administration
Drug: ropivacaine and midazolam epidural administration — Patients undergoing ACL reconstruction with hamstring autograft who will receive ropivacaine and midazolam epidural administration for anesthesic technique for the procedure
  Other Names: Ropiconest®; Ralecum®
  Arms: Ropivacaine and midazolam epidural administration

SUMMARY:
Compare of the effectiveness of the use of ropivacaine and midazolam by intraarticular vs epidural administration on post-operative analgesia after isolated arthroscopic anterior cruciate ligament (ACL) reconstruction with hamstring autograft.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) reconstruction is a common surgical knee procedure that presents moderate to severe postoperative pain, additionally, an adequate control of the pain is required to start intensive rehabilitation after the surgery, early hospital discharge and reduction of the administration of oral and intravenous anesthetic drugs.

Postoperative pain is a common upsetting symptom following ACL reconstruction that delay return to daily activity of the patient and leads to an increase in days of hospitalization and early rehabilitation.(Harris et al., 2014) Therefore, pain is also mediated by free nerve endings in the knee joint, which are located in the tendons of semitendinosus, gracilis and sartorius muscles, associated with higher pain in comparison with ACL allograft.(Hong et al., 2019) For effective, safe and longer post-ACL reconstruction analgesia, several analgesic strategies such as systemic medication, central or peripheral blocks, and intra-articular drug administration have been used to control the pain. (Baverel et al., 2016; Dauri et al., 2003; Parker et al., 2007; Peng et al., 2018; Zhou et al., 2016; Zou et al., 2016) Combined spinal anesthesia is better option for knee surgery, it can reduce the disadvantages of general and alone spinal or epidural anesthesia. Combined spinal anesthesia appears to be effective and with lower toxicity than general anesthesia. (Baldawi et al., 2020; Johnson et al., 2016; Moucha et al., 2016; Padwal et al., 2019) Moreover, reduce the hospital stay and extends the analgesia into the postoperative period without increasing morbidity. (Johnson et al., 2016)

HYPOTHESIS: The hypothesis was that there are differences in the quality and quantity of postoperative pain in knee arthroscopy surgery when midazolam plus ropivacaine is administered epidurally, in comparison to ropivacaine and midazolam by intraarticular.

Methodology:

Type of study: Controlled clinical trial. Study design: Experimental, longitudinal, comparative, prospective and double blind.

Approximate duration of the study: 12 months Population type and sample size: A total of 108 patients undergoing elective surgery for anterior cruciate ligament reconstruction after rupture Research Site: Patients will be recruited from Consultation No. 15 of the Orthopedics and Traumatology Service of the University Hospital "Dr. José Eleuterio González "of the U.A.N.L. Surgeries will be carried out in the Department of Surgical Therapeutics on the 5th floor of the University Hospital of the U.A.N.L.

Randomization mode: 108 sealed envelopes are prepared prior to the start of the study, which will include the group to which the patient will belong. The patient will not know the group to which he will belong until the moment of revealing the final results of the study.

Recruitment Methodology: Each patient who is admitted to the elective surgery of ACL reconstruction will be invited to participate voluntarily in the study. The principal investigator or one of the co-investigators will be responsible for thoroughly explaining the details of the study, including the potential benefits and risks, as well as answering any questions that may arise, if the patient agrees to participate, the patient will be asked to sign the informed consent in the presence of two witnesses and a note will be made in the clinical file where the inclusion in the study will be recorded, in the same way a copy of the consent will be given to the patient. For the purpose of the study, the identification of the patient will not be necessary only his gender, age, height and weight. The study population will be divided into 2 groups: 1. Ropivacaine plus midazolam by intra-articular application and Group 2: Ropivacaine plus midazolam epidural administration.

The surgeries of all the groups will be performed with the same surgical technique, using a total primary ACL reconstruction with TighRope ® Endobutton system. The patients will be operated by 2 subspecialists in hip joint surgery, professors of the Orthopedics and Traumatology Service of the University Hospital "Dr. José Eleuterio González "as the main surgeon and as surgical assistants to the resident doctors of Orthopedics and Traumatology.

Anesthesia protocol There were used combined spinal-epidural anesthesia. The patient was placed in lateral decubitus position. Under aseptic technique, the intervertebral space between L2-L3 or L3-L4 was superficially infiltrated with 2% lidocaine. The lumbar spinal level was identified with an 18-gauge Tuohy needle included in the spinal-epidural combined kit (Espocan®, B Braun, Germany). After that, a Whitacre 25 spinal needle was placed and the anesthesiologist confirmed the correct position by the free flow of cerebrospinal fluid. 7.5 mg (1.5 ml) of 0.5% hyperbaric bupivacaine were administered. Thereafter an epidural catheter was introduced, about 4 cm into the epidural space through the Tuohy needle for maintenance anesthesia and 60 mg (3 ml) of lidocaine with 2% epinephrine were administered to ensure the correct position outside a blood vessel. In case of prolongation of the surgical time, the anesthetic effect was extended through the epidural catheter.

Once the surgical procedure was completed and depending on the group to which the patient belongs, postoperative analgesia was administered.

Group 1. Ropivacaine with intra-articular midazolam. Ropivacaine 0.75% at 1.5 mg / kg (Ropiconest®, PiSA, Mexico) was used with midazolam at 50 mcg / kg kg (Ralecum®, PiSA, Mexico), to complete 20 ml of solution and was administrated on the knee articulation after tourniquet release. And an elastomeric pump (Home Pump® of 5 ml / hr for 24 hours) was prepared for epidural infusion, with 150 ml of physiological solution.

Group 2. Ropivacaine plus epidural midazolam. An elastomeric pump (Home Pump® of 5 ml / hr for 24 hours) was prepared for epidural infusion. This was prepared with 150 mg (20 ml) of 0.75% ropivacaine plus midazolam at 50 mcg / kg / 12 hrs. The solution was made up to 125 ml with physiological solution. Moreover, 20 ml of physiological solution, was intraarticular administered as placebo in the Ropivacaine plus epidural midazolam group.

Surgical technique All patients underwent an arthroscopic ACL reconstruction with ipsilateral hamstring autograft. There were used tourniquet in all the procedures, with the patient in supine position, with lateral positioner to perform valgus on the knee. Lateral and medial standard portals were used. A diagnostic arthroscopy was realized in all cases to check the menisci and the knee cartilage. After that the semitendinosus and gracilis tendon were harvested by a 2 cm anteromedial incision.

Repairable tears of meniscus were treated with all-inside an outside-in sutures technique. Irreparable meniscal tears were managed with partial meniscectomy and were stabilized with shaving and radio frequency cauterization of the meniscus remnant.

Drug administration protocol:

The sealed envelope will be opened on the preoperative day to identify which experimental group the patient belongs In the first group will receive an elastomeric pump was prepared for epidural infusion, with 150 ml of physiological solution and ropivacaine 0.75% at 1.5 mg / kg was used with midazolam at 50 mcg / kg kg to complete 20 ml of solution and was administrated on the knee articulation after tourniquet release.

The second group An elastomeric pump was prepared for epidural infusion. This was prepared with 150 mg (20 ml) of 0.75% ropivacaine plus midazolam at 50 mcg / kg / 12 hrs. The solution was made up to 125 ml with physiological solution. Moreover, 20 ml of physiological solution, was intraarticular administered as placebo.

The protocol for the pre and post-operative administration of the drugs will be as follows:

Only one author knew about the drugs that were administrated. The drugs were prepared in unlabeled syringes as the same volume and were recorded separately by a co-investigator who was not involved in the analysis of the study. Also, this physician, were involved in the surgery and performed anesthetic care. A blinded investigator, who was not involved in the anesthetic care of the patients, collected all study data. Surgeon, anesthesiologist and rehabilitator were blinded to group allocation.

Intrahospital follow-up Each patient was given a logbook and asked to self-evaluate and record pain (according to the 10-point VAS) before and 15 min after an analgesic administration. In case of pain with a VAS greater than 4, , 1g of acetaminophen and 30 mg IV of ketorolac were administrated. For higher than 7 points 50 mg IV of Tramadol was indicated, in any of the 2 groups, which could be repeated every 6 hours if required. In the case of the need for rescue analgesia, tramadol 50 mg IV, 30 mg IV of ketorolac and 1 g of acetaminophen were administered, the time in postoperative hours in which the first dose was administered and the total number of doses administered in 24 hours was documented, as well as the performance of equianalgesic conversion of opioids for the necessary dose used for rescue analgesia, taking into account that 200 mg IV / day of tramadol is equal to 20 mg IV / day of morphine, considered as the main reference for opioid analgesics. Tramadol 400 mg / day should not have been exceeded.

All patients who presented nausea received ondansetron 4 mg perioperative. Supplemental doses of ondansetron 1 mg were administered at the first indication of moderate to severe nausea.

Patient's discharge It will be discharged by medical indication to the patient 48 hours after surgery, if there is no type of contraindication, with indications of discharge in medical prescription and follow-up by the external consultation after one week.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years and younger than 50 years
2. Arthroscopic single bundle anterior cruciate ligament anatomic reconstruction with hamstring tendon autograft
3. Unilateral procedure
4. With or without meniscal tear
5. Desire to participate voluntarily in the study and signature of informed consent
6. Pre-operative assessment with result between (American Society of Anesthesiologist) ASA I or ASA II performed and annexed in the clinical file either by the Department of Internal Medicine, Cardiology or Anesthesiology.

Exclusion Criteria:

1. Another ligament surgery (posterior cruciate ligament, medial collateral ligament, posterolateral corner reconstruction)
2. ACL reconstruction with allograft
3. Bone to bone or quadriceps autograft
4. ACL reconstruction with double bundle technique
5. Patients with previous knee surgeries
6. Open ACL reconstruction
7. Corrective knee osteotomy or articular cartilage repair surgery, meniscal transplant, lateral extraarticular tenodesis
8. Pregnant or lactating patients
9. Patients under 18 years old
10. Patients consuming oral contraceptives
11. Patients who present any contraindication for neuraxial blockade (e.g., coagulation defects, infection at the puncture site, pre-existing neurological deficits in the lower extremities, Anticoagulant or antiplatelet therapy that has not been suspended 48 hours before the surgery, systemic infection, fever above 38.5º)
12. Preoperative assessment with ASA III-IV
13. Hypersensitivity to the drugs used in the study
14. Patients with intellectual impairments or psychiatric conditions that limited adequate communication
15. Patients with a diagnosis of fibromyalgia, polymyalgia rheumatica, complex painful syndromes or sciatic neuropathy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Post-operative analgesic request | will be measured at 24 hours after surgery
  All the medication utilized posterior to the surgery was recorded and administered in case of pain with a VAS greater than 4, the administration of 1g of acetaminophen, 30 mg IV of ketorolac and 50 mg IV of Tramadol was indicated, in any of the 2 groups, which could be repeated every 8 hours if required.

SECONDARY OUTCOMES:
Therapeutic effect on visual analog scale | Pain will be measured at 2, 6, 12 , 24 and 48 hours after surgery.
  The pain Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (scale of 10). It will be assessed as a numeric scale from 0 to 10. Being 0 better outcome than 10.
Side effects of analgesic drugs | Hemoglobin levels will be measured at 2, 6, 12 , 24 and 48 hours after surgery.]
  Focusing in sedation and postoperative nausea, measuring the need of antiemetic medication
Postoperative range of motion | at 24 and 48 hours after surgery.]
  Measured in the grades of flexion and extension after surgery
Post-operative analgesic request | will be measured at 2, 6, 12 , 24 and 48 hours after surgery.
  All the medication utilized posterior to the surgery was recorded and administered in case of pain with a VAS greater than 4, the administration of 1g of acetaminophen, 30 mg IV of ketorolac and 50 mg IV of Tramadol was indicated, in any of the 2 groups, which could be repeated every 8 hours if required.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Morales-Avalos, MSc, MD, Principal Investigator — University Hospital "Dr. José Eleuterio González", Universidad Autonoma de Nuevo León (U.A.N.L.)
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Result] Baldawi M, McKelvey G, Saasouh W, Perov S, Mostafa G, Saleh K. A Comparison of Neuraxial and General Anesthesia for Thirty-Day Postoperative Outcomes in United States Veterans Undergoing Total Knee Arthroplasty. J Arthroplasty. 2020 Nov;35(11):3138-3144. doi: 10.1016/j.arth.2020.06.030. Epub 2020 Jun 17. PMID 32641270
- [Result] Baverel L, Cucurulo T, Lutz C, Colombet, Cournapeau J, Dalmay F, Lefevre N, Letartre R, Potel JF, Roussignol X, Surdeau L, Servien E; French Arthroscopic Society. Anesthesia and analgesia methods for outpatient anterior cruciate ligament reconstruction. Orthop Traumatol Surg Res. 2016 Dec;102(8S):S251-S255. doi: 10.1016/j.otsr.2016.08.007. Epub 2016 Sep 26. PMID 27687059
- [Result] Dauri M, Polzoni M, Fabbi E, Sidiropoulou T, Servetti S, Coniglione F, Mariani P, Sabato AF. Comparison of epidural, continuous femoral block and intraarticular analgesia after anterior cruciate ligament reconstruction. Acta Anaesthesiol Scand. 2003 Jan;47(1):20-5. doi: 10.1034/j.1399-6576.2003.470104.x. PMID 12492792
- [Result] Hong AJ, Agarwalla A, Liu JN, Gowd AK, McMillan S, Sethi PM, Amin NH. Neurological structures and mediators of pain sensation in anterior cruciate ligament reconstruction. Ann Anat. 2019 Sep;225:28-32. doi: 10.1016/j.aanat.2019.05.010. Epub 2019 Jun 11. PMID 31195095
- [Result] Johnson RL, Kopp SL, Burkle CM, Duncan CM, Jacob AK, Erwin PJ, Murad MH, Mantilla CB. Neuraxial vs general anaesthesia for total hip and total knee arthroplasty: a systematic review of comparative-effectiveness research. Br J Anaesth. 2016 Feb;116(2):163-76. doi: 10.1093/bja/aev455. PMID 26787787
- [Result] Lauretti GR, de Oliveira R, Perez MV, Paccola CA. Postoperative analgesia by intraarticular and epidural neostigmine following knee surgery. J Clin Anesth. 2000 Sep;12(6):444-8. doi: 10.1016/s0952-8180(00)00189-6. PMID 11090729
- [Result] Nahravani M, Tekye SM, Alipour M, Makhmalbaf H, Aghaee MA. Analgesia Following Arthroscopy - a Comparison of Intra-articular Bupivacaine and/or Midazolam and or Fentanyl. Arch Bone Jt Surg. 2017 Jan;5(1):28-31. PMID 28271084
- [Result] Padwal JA, Burton BN, Fiallo AA, Swisher MW, Gabriel RA. The association of neuraxial versus general anesthesia with inpatient admission following arthroscopic knee surgery. J Clin Anesth. 2019 Sep;56:145-150. doi: 10.1016/j.jclinane.2019.01.045. Epub 2019 Feb 23. PMID 30807886
- [Result] Parker RD, Streem K, Schmitz L, Martineau PA; Marguerite Group. Efficacy of continuous intra-articular bupivacaine infusion for postoperative analgesia after anterior cruciate ligament reconstruction: a double-blinded, placebo-controlled, prospective, and randomized study. Am J Sports Med. 2007 Apr;35(4):531-6. doi: 10.1177/0363546506296313. Epub 2007 Jan 23. PMID 17244900
- [Result] Peng K, Chen WR, Meng XW, Zhang J, Ji FH. Intra-articular dexmedetomidine in knee arthroscopy: A systematic review and meta-analysis. Sci Rep. 2018 Mar 6;8(1):4089. doi: 10.1038/s41598-018-22482-8. PMID 29511256
- [Result] Zhou Y, Yang TB, Wei J, Zeng C, Li H, Yang T, Lei GH. Single-dose intra-articular ropivacaine after arthroscopic knee surgery decreases post-operative pain without increasing side effects: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1651-9. doi: 10.1007/s00167-015-3656-y. Epub 2015 Jun 7. PMID 26049805
- [Result] Zou Z, An MM, Xie Q, Chen XY, Zhang H, Liu GJ, Shi XY. Single dose intra-articular morphine for pain control after knee arthroscopy. Cochrane Database Syst Rev. 2016 May 3;2016(5):CD008918. doi: 10.1002/14651858.CD008918.pub2. PMID 27140500